CLINICAL TRIAL: NCT05930925
Title: AN INTERVENTIONAL, PHASE 1, OPEN-LABEL, 2-ARM PARALLEL STUDY TO INVESTIGATE THE ABSORPTION, METABOLISM, AND EXCRETION OF [14C]ARV-471 IN HEALTHY ADULT PARTICIPANTS
Brief Title: A Study to Understand How the Study Medicine Called ARV-471 is Processed in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Arvinas Estrogen Receptor, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: C4891014
Record Dates: First submitted 2023-06-08; First posted 2023-07-05 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- [phenyl-14C]ARV-471 (Experimental): [phenyl-14C]ARV-471 is administered as a single dose
  Interventions: Drug: [phenyl-14C]ARV-471
- [oxoisoindolin-14C]ARV-471 (Experimental): [oxoisoindolin-14C]ARV-471 is administered as a single dose
  Interventions: Drug: [oxoisoindolin-14C]ARV-471

INTERVENTIONS:
Drug: [phenyl-14C]ARV-471 — Participants will receive a single dose of [phenyl-14C]ARV-471 by mouth
  Arms: [phenyl-14C]ARV-471
Drug: [oxoisoindolin-14C]ARV-471 — Participants will receive a single dose of [oxoisoindolin-14C]ARV-471 by mouth
  Arms: [oxoisoindolin-14C]ARV-471

SUMMARY:
The purpose of the study is to understand how the study medicine ARV-471 is processed in the body of healthy males and females who do not have the potential to have children.

This study is seeking for participants who:

* are healthy males and females who do not have the potential to have children.
* are 18 years of age or older.
* weigh more than 110 pounds.

DETAILED DESCRIPTION:
About 6 participants each will receive a single dose of either type of ARV-471. They are taken as liquid suspensions by mouth. Participants will stay in the study site for about 13 days and 12 nights.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 18 years or older (or the minimum age of consent in accordance with local regulations) at screening.
* Male and female participants of non-childbearing potential who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and ECG monitoring.
* Total body weight >50 kg (110 lb).
* An informed consent document signed and dated by the subject.
* Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).

  * Any condition possibly affecting drug absorption (eg, gastrectomy, cholecystectomy).
  * History of clinically significant thromboembolic or cerebrovascular events.
  * History of HIV infection, hepatitis B, or hepatitis C; positive testing for HIV, HBsAg, or HCVAb. Hepatitis B vaccination is allowed.
* Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
* Use of prescription or nonprescription medications, including vitamins, dietary and herbal supplements are prohibited in this study. A washout of 7 days or 5 half-lives (whichever is longer) prior to the first dose of study intervention is required, or a longer washout is required for those that fall into the categories below:

  * Moderate/strong CYP3A inducers; these are prohibited within 14 days plus 5 half-lives prior to the first dose of study intervention.
  * Moderate/strong CYP3A inhibitors; these are prohibited within 14 days or 5 half lives (whichever is longer) prior to the first dose of study intervention.
* Previous administration with an investigational product (drug or vaccine) within 30 days (or as determined by the local requirement) or 5 half lives preceding the first dose of study intervention used in this study (whichever is longer).
* A positive urine drug test.
* Screening supine BP ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic), following at least 5 minutes of supine rest.
* Renal impairment as defined by an eGFR in adults of <60 mL/min.
* Hematuria as defined as >1+ heme on urine dipstick.
* Proteinuria or Albuminuria as defined as >1+ protein on urine dipstick OR positive dipstick for albumin OR Albumin/Cr ratio on spot urine (UA) >30 mg/g.
* Standard 12 lead ECG that demonstrates clinically relevant abnormalities that may affect participant safety or interpretation of study results (eg, QTcF >450 ms, complete LBBB, signs of an acute or indeterminate age myocardial infarction, ST T interval changes suggestive of myocardial ischemia, second- or third-degree AV block, or serious bradyarrhythmias or tachyarrhythmias).
* Participants with ANY of the following abnormalities in clinical laboratory tests at screening, as assessed by the study specific laboratory and confirmed by a single repeat test, if deemed necessary:

  * AST or ALT level >1.0× ULN;
  * Total bilirubin level >1.0 × ULN; participants with a history of Gilbert's syndrome may have direct bilirubin measured and would be eligible for this study provided the direct bilirubin level is ≤ ULN.
* History of alcohol abuse or binge drinking and/or any other illicit drug use or dependence within 6 months of Screening. Binge drinking is defined as a pattern of 5 (male) and 4 (female) or more alcoholic drinks in about 2 hours. As a general rule, alcohol intake should not exceed 14 units per week (1 unit = 8 ounces (240 mL) beer, 1 ounce (30 mL) of 40% spirit, or 3 ounces (90 mL) of wine).
* Blood donation (excluding plasma donations) of approximately 1 pint (500 mL) or more within 60 days prior to dosing.
* History of sensitivity to heparin or heparin induced thrombocytopenia.
* Unwilling or unable to comply with the criteria in the Lifestyle Considerations section of this protocol.
* Investigator site staff directly involved in the conduct of the study and their family members, site staff otherwise supervised by the investigator, and sponsor and sponsor delegate employees directly involved in the conduct of the study and their family members.
* History of sensitivity to ARV-471 or any of the formulation components of ARV 471.
* Participants with a history of irregular bowel movements (eg, regular episodes of diarrhea or constipation, or IBS).
* Participants enrolled in a previous radionucleotide study or who have received radiotherapy within 12 months prior to screening or such that total radioactivity would exceed acceptable dosimetry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-06-12 (Actual); Primary Completion 2023-07-27 (Actual); Study Completion 2023-08-14 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - ∞)] of ARV-471 and ARV-473 (an epimer of ARV-471) | Day 1 pre-dose, 1, 2, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, 144, 168, 192, 216, 240, 264 hours post-dose
Maximum Observed Plasma Concentration (Cmax) of ARV-471 and ARV-473 (an epimer of ARV-471) | Day 1 pre-dose, 1, 2, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, 144, 168, 192, 216, 240, 264 hours post-dose
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) of ARV-471 and ARV-473 (an epimer of ARV-471) | Day 1 pre-dose, 1, 2, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, 144, 168, 192, 216, 240, 264 hours post-dose
Time to Reach Maximum Observed Plasma Concentration (Tmax) of ARV-471 and ARV-473 (an epimer of ARV-471) | Day 1 pre-dose, 1, 2, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, 144, 168, 192, 216, 240, 264 hours post-dose
Plasma Decay Half-Life (t1/2) of ARV-471 and ARV-473 (an epimer of ARV-471) | Day 1 pre-dose, 1, 2, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, 144, 168, 192, 216, 240, 264 hours post-dose
Apparent Oral Clearance (CL/F) of ARV-471 | Day 1 pre-dose, 1, 2, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, 144, 168, 192, 216, 240, 264 hours post-dose
Apparent Volume of Distribution (Vz/F) of ARV-471 | Day 1 pre-dose, 1, 2, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, 144, 168, 192, 216, 240, 264 hours post-dose
Renal Clearance (CLr) of ARV-471 and ARV-473 (an epimer of ARV-471) | Day 1 at intervals of 0-6 hours, 6-12 hours, 12-24 hours, and at each subsequent 24-hour interval starting on Day 2 until Day 12 or the discharge day
Cumulative Amount of Drug Recovered Unchanged in Urine (Ae) of ARV-471 and ARV-473 (an epimer of ARV-471) and the Total Amounts Expressed as a Percent of Dose (Ae(%)) | Day 1 at intervals of 0-6 hours, 6-12 hours, 12-24 hours, and at each subsequent 24-hour interval starting on Day 2 until Day 12 or the discharge day
Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - ∞)] of Total Radioactivity | Day 1 pre-dose, 1, 2, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, 144, 168, 192, 216, 240, 264 hours post-dose
Maximum Observed Plasma Concentration (Cmax) of Total Radioactivity | Day 1 pre-dose, 1, 2, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, 144, 168, 192, 216, 240, 264 hours post-dose
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) of Total Radioactivity | Day 1 pre-dose, 1, 2, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, 144, 168, 192, 216, 240, 264 hours post-dose
Time to Reach Maximum Observed Plasma Concentration (Tmax) of Total Radioactivity | Day 1 pre-dose, 1, 2, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, 144, 168, 192, 216, 240, 264 hours post-dose
Plasma Decay Half-Life (t1/2) of Total Radioactivity | Day 1 pre-dose, 1, 2, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, 144, 168, 192, 216, 240, 264 hours post-dose
Apparent Oral Clearance (CL/F) of Total Radioactivity | Day 1 pre-dose, 1, 2, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, 144, 168, 192, 216, 240, 264 hours post-dose
Apparent Volume of Distribution (Vz/F) of Total Radioactivity | Day 1 pre-dose, 1, 2, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, 144, 168, 192, 216, 240, 264 hours post-dose
Cumulative recovery (%) of radioactivity in urine and feces | Starting on Day 1 to Day 12 or the discharge day
Metabolite identification/profiling in feces, plasma and urine | Day 1 pre-dose, 1, 2, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, 144, 168, 192, 216, 240, 264 hours post-dose

SECONDARY OUTCOMES:
Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs) | Time the participant provides informed consent through and including follow-up contact occurring 28 to 35 calendar days after the last administration of the study intervention.
  An AE is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship with the study treatment. SAE is defined as one of the following: is fatal or life-threatening; results in persistent or significant disability/incapacity; constitutes a congenital anomaly/birth defect; is medically significant; requires inpatient hospitalization or prolongation of existing hospitalization. Treatment-emergent AE is defined as an AE with onset date occurring during the on-treatment period. AEs include all SAEs and non-SAEs.
Number of Participants With Clinical Laboratory Abnormalities | Baseline up to Day 12/Discharge
  Following parameters were analyzed for laboratory examination: hematology(hemoglobin, hematocrit, red blood cell count, platelet count, white blood cell count, total neutrophils, eosinophils, monocytes, basophils, lymphocytes); liver function(aspartate aminotransferase, alanine aminotransferase, total bilirubin, alkaline phosphatase, albumin, total protein); renal function (blood urea nitrogen, creatinine, uric acid, cystatin C);electrolytes (sodium, potassium, chloride, calcium, bicarbonate); clinical chemistry(glucose); urinalysis (dipstick[decimal logarithm of reciprocal of hydrogen ion activity {pH} of urine, glucose, protein, blood, ketones, nitrites, leukocyte esterase, urobilinogen, bilirubin], microscopy.
Number of Participants With Electrocardiogram (ECG) Abnormalities | Baseline up to Day 12/Discharge
  ECG abnormalities criteria include a) a post dose QTcF is increased by >60 ms from the baseline and is >450 ms; or b) an absolute QTcF value is >500ms for any scheduled ECG.
Number of Participants With Clinically Significant Change From Baseline in Vital Signs | Baseline up to Day 12/Discharge
  Blood pressure and pulse rate will be performed following at least a 5-minute rest in a supine position.
Number of Participants With Abnormalities in Physical Examinations | Baseline up to Day 12/Discharge
  A complete physical examination will include, at a minimum, head, ears, eyes, nose, mouth, skin, heart and lung examinations, lymph nodes, and gastrointestinal, musculoskeletal, and neurological systems.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- PPD Phase I Clinic, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4891014